CLINICAL TRIAL: NCT06935916
Title: Retrospective Analysis of Surgical Outcomes in Patients Treated for Gunshot-Related Bone Defects at Mekelle University Hospital
Status: Completed | Type: Observational
Sponsor: Julian Joestl (Other)
Responsible Party: Sponsor-Investigator, Julian Joestl, Clinical Professor PD DDr. MSc., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: GSR/0832/10
Record Dates: First submitted 2025-04-06; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Reconstructive Surgery
Keywords: free fibula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who underwent pedicled or free tissue transfer: patients who underwent pedicled or free tissue transfer
  Interventions: Procedure: pedicled or free tissue transfer

INTERVENTIONS:
Procedure: pedicled or free tissue transfer — pedicled or free tissue transfer

SUMMARY:
his project looks back at past surgeries performed between 2019 and 2023 in a hospital in Mekelle, Ethiopia. During this time, a team of doctors from Austria and other countries visited the hospital to help patients who had been badly injured by gunshots, especially in the legs and arms. These injuries were very serious and often needed complex operations.

Why is this important? Mekelle is in a region that was affected by conflict and war. Hospitals there have very limited resources - not enough electricity, medical tools, or staff. The patients are often young people with injuries that would be easier to treat in better-equipped hospitals. This project wants to understand how the surgeries went under these difficult conditions and what could be done better in the future.

What will the doctors do in this study? They will look at hospital records from about 74 patients who had these surgeries. The doctors will not contact patients or do any new treatments. They are only using data that was already collected during treatment. The names and personal details of patients will not be used - everything will be anonymous.

The doctors will study:

The age and gender of patients What type of surgery was done How long surgeries lasted and whether electricity was available What happened after surgery - for example, whether the wound healed well or if there were problems What is the goal? The goal is to learn what worked well and what didn't - and to use this knowledge to plan future humanitarian missions. The results could also help improve care for people in similar situations in other parts of the world.

Are there any risks? No. This is a purely retrospective study. That means it only looks at past data. There will be no contact with patients, and no further action taken based on the study. All personal information will be protected according to strict privacy rules.

Who is behind this project? The project is led by Dr. Viktoria Koenig, a plastic surgeon from Austria who took part in the missions and has experience with this kind of surgery.

Why is this relevant? This study will help medical teams better prepare for working in difficult environments. It will also show how surgery can still help people even when resources are very limited - and highlight the importance of teamwork, planning, and flexible medical approaches.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent pedicled or free tissue transfer during the study period

Exclusion Criteria:

* All other patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent pedicled or free tissue transfer during the study period
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Survival rate of the transferred tissue | Perioperative/Periprocedural
  Survival rate of the transferred tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Medical university of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gufue ZH, Haftu HK, Alemayehu Y, Tsegay EW, Mengesha MB, Dessalegn B. Damage to the public health system caused by war-related looting or vandalism in the Tigray region of Northern Ethiopia. Front Public Health. 2024 Apr 5;12:1271028. doi: 10.3389/fpubh.2024.1271028. eCollection 2024. PMID 38645448